CLINICAL TRIAL: NCT06834022
Title: Comparison of Neuromodulatory Treatment of Migraine Headache with Acupuncture and Transcranial Direct Current Stimulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Alenka Spindler-Vesel, MD, PhD, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0120-421/2022/3
Record Dates: First submitted 2023-05-11; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Migraine
Keywords: tDCS; acupuncture; CGRP; inflammatory biomarkers
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Direct Current Stimulation; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sham Acupuncture (Placebo Comparator): Patients receive sham acupuncture (skin remains intact, away from standard acupuncture points)
  Interventions: Procedure: Acupuncture
- Verus Acupuncture (Active Comparator): Patients receive acupuncture treatment over semistandardized acupuncture points for migraine headache.
  Interventions: Procedure: Acupuncture
- Sham tDCS (Placebo Comparator): Device will provide only placebo stimulation (study mode)
  Interventions: Device: Transcranial direct current stimulation
- verus tDCS (Active Comparator): Device will stimulate with direct current (study mode)
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS will be used according to instructions for use in migraine headache (supraorbital and M1 stimulation), 1 mA, 20 min, 10 sessions
  Arms: Sham tDCS; verus tDCS
Procedure: Acupuncture — Acupuncture will be semistandardized, (every patient is stimulated over Li4, St36, Li3 + patient specific acu-points), 10 sessions
  Arms: Sham Acupuncture; Verus Acupuncture

SUMMARY:
The goal of this clinical trial is to compare effects of the treatment with acupuncture and transcranial direct current stimulation (tDCS) in patients with migraine headache. The main questions it aims to answer are:

* is tDCS more effective than acupuncture/placebo?
* is there any difference in venous blood inflammatory parameters (CGRP (calcitonin gene related peptide), IL (interleukine) -6, IL-8. IL-10, SAA (serum amyloid A) and ESR (erythrocyte sedimentation rate) before/after treatment?
* could these inflammatory parameters function as biomarkers of disease and/or indicators of treatment's efficacy?

Participants will regularly fill out questionnaires (migraine diary) and their venous blood before/after treatment will be taken for analysis.

Researchers will compare the effects of sham and verus treatment of both methods before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 4 migraine days per month
* no acupuncture in the past
* understanding of study design and ability to give informed consent

Exclusion Criteria:

* severe psychiatric disorders
* pacemaker
* status post brain surgery with open skull
* brain stimulators
* metal implants
* biologic drugs
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of days with migraine headache per month | 4 months
  Evaluation of migraine days before study, at 1 nad 3 months after comleted therapy.

SECONDARY OUTCOMES:
Severity of migraine headache | 4 months
  Evaluation of HIT and MIDAS questionnaire before study and 1 and 3 months after completed therapy.
  CGRP levels before and after 1 and 3 months after completed therapy
Change of inflammatory parameters | 4 months
  Measurements of laboratory levels of IL-6, IL-8, IL-10, leptin before treatment and at 1 and 3 months after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Manja Mlakar, MD, Principal Investigator — University of Ljubljana
Locations (1):
- Hospital dr. Petra Držaja, Ljubljana, Ljubljana, Slovenia